CLINICAL TRIAL: NCT04105283
Title: Tc99m-MAA Bronchial Artery Injection During Bronchial Embolization for Pulmonary Mass Induced Hemoptysis for Dosimetry Planning
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: BTG International Inc. (Other)
Responsible Party: Principal Investigator, Eric Wehrenberg-Klee, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-218
Record Dates: First submitted 2019-09-20; First posted 2019-09-26 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Technetium Tc 99m Aggregated Albumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tc99m-MAA (Experimental): * Tc99m-MAA will be administered by selective or supra-selective arterial injection via the bronchial artery or branches thereof.
  * Administration will occur over a period of 30-240 seconds
  Interventions: Biological: Tc99m-MAA

INTERVENTIONS:
Biological: Tc99m-MAA — Tc99m-MAA is a particle that is used to assess blood flow distribution and has a similar size to the particles that are utilized for arterial delivery of radiation therapy, also called radioembolization. Tc99m-MAA is currently used to estimate radiation dosimetry prior to arterial radiotherapy administration for liver malignancies.

SUMMARY:
This research study will evaluate the administration of a particle called macro-aggregated albumin (MAA) labelled with the radiotracer technetium 99m (Tc99m) as a proxy to estimate the anticipated dose of radiation to tumor and adjacent structures.

Administration of this labeled MAA will not have a therapeutic benefit on the participant's cancer. Administration will help researchers determine if arterial administration of radiation may be feasible for lung cancer in the future.

DETAILED DESCRIPTION:
This research study is a Pilot Study, which is the first time investigators are examining this study intervention.

As mentioned above, standard of care treatment for Stage III lung cancer includes chemotherapy and stereotactic body radiation therapy. However, arterial administration of radiation to these tumors may represent an alternative method of radiotherapy, with dose directly administered to the tumor. The potential radiation dose to the tumor and adjacent structures is not known.

This study aims to estimate the dose of radiation to tumor and adjacent structures in the chest via administration of a radiotracer called Tc99m-MAA. Tc99m-MAA is a particle that is used to assess blood flow distribution and has a similar size to the particles that are utilized for arterial delivery of radiation therapy, also called radioembolization. Tc99m-MAA is currently used to estimate radiation dosimetry prior to arterial radiotherapy administration for liver malignancies.

If this study is successful, the results will allow doctors to use the distribution of Tc99m-MAA to estimate radiation dose to tumors and adjacent structures in the setting of intra-arterial radiation therapy. This will provide information to plan future therapy with intra-arterial radioembolization for lung malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age and older
* Patients with known active lung cancer with a history of hemoptysis presenting for standard of care bronchial artery embolization will be considered.
* Patients must be presenting for secondary prophylaxis of hemoptysis.
* If female, not of childbearing potential or negative serum β-hCG pregnancy test prior to CTA chest and radiotracer injection.
* If female, not nursing.
* Willing and able to understand and sign a written informed consent document.
* Willing and able to undergo all study procedures

Exclusion Criteria:

* Patients with current active hemoptysis
* Any acute or chronic inflammatory disease or medical conditions that in the investigator's opinion may interfere with the study procedures or the interpretation of the study results.
* Subjects who have exclusion criteria that would prevent them from receiving a CT scan or fluoroscopy, or administration of contrast.
* History of allergic reactions or hypersensitivity attributed to compounds of similar chemical or biologic composition to macro-aggregated albumin
* Patients with severe pulmonary hypertension.
* Glomerular filtration rate < 30
* Platelets < 30
* INR > 3.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Calculation of Tc99m-MAA uptake within the tumor and surrounding structures (radioactivity concentration) | 2 years

SECONDARY OUTCOMES:
Number of patients experiencing off-target administration of Tc99m-MAA to distant organs (as assessed by radioactivity concentration assessed in regions of interest in distant extremities, head, abdomen) | 2 years
Number of patients experiencing immediate post-procedural adverse events associated with bronchial artery administration of Tc99m-MAA | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wehrenberg-Klee, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation
URL: http://www.partners.org/innovation

REFERENCES:
- [Derived] Wehrenberg-Klee E, An T, Heidari P, Huesa-Berral C, Dreher MR, Eldridge A, Fowers K, Schuemann J, Bertolet A. SPECT/CT Dosimetry of Bronchial Artery 99mTc Macroaggregated Albumin Injection in Pulmonary Malignancies: Feasibility Evaluation of Bronchial Artery 90Y Radioembolization. Radiology. 2025 Feb;314(2):e240331. doi: 10.1148/radiol.240331. PMID 39964268